CLINICAL TRIAL: NCT04531683
Title: Efficacy and Safety of Electroacupuncture on Mixed Urinary Incontinence Among Women: a Multi-centre, Randomised Controlled Trial
Brief Title: Effect of Electroacupuncture on Mixed Urinary Incontinence Among Women
Acronym: EAMUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Shaanxi Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Heilongjiang University of Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Chief Physician, Dean of Acupuncture Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZZ13-024-9
Record Dates: First submitted 2020-08-20; First posted 2020-08-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence, Mixed
Keywords: acupuncture; randomised controlled trial; sham acupuncture
MeSH Terms: conditions — Urinary Incontinence | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Patients who sign the informed consent form and are eligible for the study entry at week 0 will be randomised to one of the three groups: electro-acupuncture group, sham electroacupuncture group and life style consultation group. The three group will be assessed in a paralleled manner, and patients in the first two groups will be treated 3 times per week for 8 weeks and followed up for 24 weeks, while patients in the third group will be provided with life style improvement information once and followed-up for 20 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigator and outcome assessor will be masked. The care provider will be different from investigator and outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture (Experimental): patients will receive electroacupuncture at 3 acupoints (Bladder meridian of foot-taiyang 33 and 35（BL33 and BL35), and Spleen meridian of foot-taiyin 33(SP6)) 3 times/week for 8 weeks(24 times in total), followed with 24-weeks follow up. Disposable acupuncture needles with size of 0.30 × 75 mm will be used at BL 33 and BL 35, and needles with size of 0.30 × 40 mm at SP 6. Standardised electroacupuncture apparatuses will be used, and the stimulation will last for 30 minutes with a continuous wave of 20 Hz, and a current intensity of 2 to 6.5 mA at BL33 and BL 35, and 1 to 3.5 mA at SP6. Life style counselling will be provided to all patients and contents are as same as the life style counselling group.
  Interventions: Other: electroacupuncture; Behavioral: life style counselling
- sham electroacupuncture (Sham Comparator): patient will receive sham electroacupuncture with the same frequency and amount as applied in the electroacupuncture group, as well as the follow-up period. Disposable acupuncture needles with size of 0.30 × 40 mm will be applied and penetrate the skin of patients for 2 to 3mm at sham acupoints to the 3 acupoints mentioned above. The stimulation will only last for 30-second with a very weak currency intensity and a continuous wave of 20 Hz. Life style counselling will be provided to all patients and contents are as same as the life style counselling group.
  Interventions: Other: sham electroacupuncture; Behavioral: life style counselling
- life style counselling group (Other): patients randomised to this group will receive a one-time life style counselling at the enrolment to improve their daily behaviour to expedite the recovery of their mixed urinary incontinence. Then the patients will be followed up for 20 weeks.
  Interventions: Behavioral: life style counselling

INTERVENTIONS:
Other: electroacupuncture — same as described in experimental arm.
  Arms: electroacupuncture
Other: sham electroacupuncture — same as described in sham comparator.
  Arms: sham electroacupuncture
Behavioral: life style counselling — life style counselling to patients with mixed urinary incontinence contains advice on daily drinking, caffeine intake, diet, constipation, exercise, heavy lifting, lung disease, urinary track infection and etc.

SUMMARY:
The purpose of the study is to assess the efficacy and safety of electroacupuncture on mixed urinary incontinence among women.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent form will be undergo a 1-week screening period to determine eligibility for study entry. Eligible patients will be randomly assigned to one of the three groups 1) electroacupuncture group: electroacupuncture will be provided to patients at BL33, BL35 and SP6 for 3 time per week for 8 weeks; 2) sham electroacupuncture group: sham electroacupuncture will be provided to patients at sham acupoints to BL33, BL35 and SP6 for 3 time per week for 8 weeks.The follow-up time for the first two groups are 24 weeks and life style counselling will be provided once when receiving the first acupuncture treatment(contents are the same as the life style counselling group). 3) life style counselling group: life style advice will be provided to patients at enrolment with content on drinking, diet, weight control, lung disease, urinary track infection control, and etc. Patients in this group will be followed up for 20 weeks. Primary and secondary outcome will be measured at 4, 8, 20, 32 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are female and meet the diagnosis criteria of mixed urinary incontinence;
2. Patients are between age of 35 to 75 years old;
3. Positive in cough stress test;
4. Experience persistent urinary incontinence for at least 3 months, and at least one episode for each of stress and urgent urinary incontinence in 72 hours in baseline screening; and
5. Patients have signed informed consent form and are willing to participate the study voluntarily.

Patients will be included if all above 5 items are met.

Exclusion criteria:

1. Patients have simple stress urinary incontinence, simple urgent urinary incontinence, overflowing urinary incontinence and neurogenic bladder, etc.;
2. Patients have uncontrolled urinary tract infection with urinary pain and urge;
3. Patients have urogenital system tumours and/or pelvic organ tumours;
4. Patients have taken drugs for urinary incontinence treatment or drugs possibly affect the function of lower urinary tract, or received non-drug treatment for urinary incontinence (i.e. electrical stimulation, bladder training, pelvic floor muscle training, and etc.) in the past one month;
5. Patients have history of surgeries for urinary incontinence and/or pelvic floor organs, including hysterectomy;
6. Patients have pelvic organ prolapse ≥ II degree;
7. Patients have residual urine ≥ 100ml;
8. Patients have uncontrolled diabetes mellitus and severe hypertension;
9. Patients have diseases affecting lower urinary tract function, e.g. multiple sclerosis, Alzheimer's disease, Parkinson's disease, spinal cord injury, cauda equina injury and multiple system atrophy, etc.;
10. Patients have severe heart, lung, brain, liver, kidney and hematopoietic system diseases, mental disorders and cognitive dysfunction;
11. Patients are constrained or unable to complete movements like walking, going stairs up and down and running, etc.;
12. Patients have poor compliance;
13. Patients are at pregnancy, breastfeeding or postpartum period for less than 12 months;
14. Patients have cardiac pacemaker, metal allergy or strong fear of needle;
15. Patients are participants of other on-going studies; or
16. Patients have received acupuncture in the past 3 months. Patients will be excluded if they meet any of the above criteria.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour incontinence episodes. | at the 8th week after the last treatment
  data will be collected and evaluated by 72-hour incontinence episodes dairy

SECONDARY OUTCOMES:
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour incontinence episodes | at baseline, 4th, 20th and 32nd week
  data will be collected and evaluated by 72-hour incontinence episodes dairy
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour urgent incontinence episodes | at baseline, 4th, 8th 20th and 32nd week
  data will be collected and evaluated by 72-hour incontinence episodes dairy
the proportion of participants with at least 50 percent decrease from baseline in the mean 24-hour stress incontinence episodes | at baseline, 4th, 8th, 20th and 32nd week
  data will be collected and evaluated by 72-hour incontinence episodes dairy
the change from baseline in the amount of urine leakage measured by the 1-hour pad test | at baseline, and the 8th week
  data will be collected by 1-hour pad test
the change from baseline in the validated Chinese version of International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF) scores | at baseline, 4th, 8th, 20th and 32nd week
  data will be collected via International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF). The total score(0-21scores) is an accumulated scores from question 1 to 3. The higher the total score is, the severer the incontinence is.
the change from baseline in the validated Chinese version of the Overactive Bladder Questionnaire-Short Form scores | at baseline 4th, 8th, 20th and 32nd week
  data will be collected via the Overactive Bladder Questionnaire-Short Form. The higher the total score is, the severer the condition is.
number of patients with one or more life style change | at the 4th, 8th, 20th and 32nd week
  life style change, such as drinking, diet, weight control and etc, will be evaluated through questionnaire
incidence rate of any adverse events | this is a case-based data reported by each centre from the start of treatment to the end of follow-up, up to 1 year and 4 months.
  adverse event associated either with or without acupuncture will be documented as soon as it is reported in any centres. The type of conditions, time of on-set and relief, its relation with the intervention, treatment to the adverse event, whether the patient's participation is terminated or not due to the adverse event, etc.
patients' expectation to treatment | at baseline
  patients will be asked about their expected effect of the treatment via question: In your expectation, how is your incontinence like in a two month time. Five choices will be provided 1) much better; 2) slightly better; 3) I don't know; 4) no change; 5) worse.
blinding assessment | in 8th week after any acupuncture treatment
  patients will be asked whether they received electroacupuncture or sham acupuncture to assess the effect of blinding

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No
We cannot share IPD under current regulation of Human Genetic Resources Management in China.